CLINICAL TRIAL: NCT05724342
Title: Tenecteplase REperfusion in Acute Ischemic sTroke Registry
Brief Title: Tenecteplase REperfusion in Acute Ischemic sTroke Registry（TREAT）
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Beijing Municipal Science & Technology Commission (Other); Beijing Municipal Administration of Hospitals (Other Government)
Responsible Party: Principal Investigator, Yunyun Xiong, Professor of Neurology and Stroke Center, Beijing Tiantan Hospital
Other Study IDs: KY2022-236-02
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Stroke, Ischemic
Keywords: thrombolysis; tenecteplase
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- rhTNK-tPA Thrombolysis
  Interventions: Drug: rhTNK-tPA Thrombolysis

INTERVENTIONS:
Drug: rhTNK-tPA Thrombolysis — rhTNK-tPA Thrombolysis

SUMMARY:
The aim of the study was to establish tenecteplase thrombolysis database and to investigate the effectiveness and safety of rhTNK-tPA in acute ischemic stroke patients.

DETAILED DESCRIPTION:
Tenecteplase (TNK), as a newer fibrinolytic agent, has practical delivery advantages over alteplase that would make it a potential alternative. Several randomized controlled clinical trials demonstrated the noninferiority of TNK but the evidence on the effectiveness and safety of TNK in the real-world is insufficient.

This is a multi-center, prospective, registry cohort study that enrolled acute ischemic stroke patients treated with TNK thrombolysis in China.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years;
* Diagnosed as acute ischemic stroke；
* Time intervals ≤ 4.5 hours from stroke onset to thrombolysis with TNK(Perfusion imaging completed including CTA+CTP or MRA+PWI+DWI before thrombolysis if the time intervals from stroke onset to thrombolysis was ≥4.5 hours)；
* Thrombolysis with rhTNK-tPA and derivatives.

Exclusion Criteria:

* Unlikely to adhere to the study protocol or follow-up ( life expectancy ≤ 3 months)；
* Already participated in other interventional trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute ischemic stroke patients treated with rhTNK-tPA and derivatives in China.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Excellent functional outcome at 90 days | 3 months after thrombolysis
  proportion of mRS score 0-1 at 3 months. The modified Rankin Scale (mRS) has a minimum value of 0 and maximum value of 6. Higher value indicated worse functional outcome

SECONDARY OUTCOMES:
Favorable functional outcome | 3 months after thrombolysis
  proportion of mRS score 0-2 at 3 months
Walk independence | 3 months after thrombolysis
  proportion of mRS score 0-3 at 3 months
Ordinal distribution of mRS at 90 days | 3 months after thrombolysis
  Number of participants with the ordinal distribution of mRS at 90 days
Neurological improvement at 24 hours | 24 hours after thrombolysis
  NIHSS score <=1 or improvement of NIHSS score>=4 compared with baseline NIHSS. National Institution Health Stroke Scale (NIHSS) has a minimum value of 0 and maximum value of 45. Higher value indicated worse severity of neurological impairment.
NIHSS score at discharge | 5-7days after thrombolysis or at discharge
  NIHSS score at 5-7 days or at discharge
EQ-5D score at 90 days | 3 months after thrombolysis
  EQ-5D score at 3 months. EuroQol Five Dimensions Questionnaire scale (EQ-5D score) has a minimum value of 0 and maximum value of 100. Lower value indicated worse functional outcome
Barthel(BI) at 90 days | 3 months after thrombolysis
  Global function of daily living defined as BI ≥ 95 at 90 days

OTHER OUTCOMES:
Symptomatic intracerebral hemorrhage at 36 hours | 36 hours after thrombolysis
  symptomatic intracerebral hemorrhage as defined by ECASSIII: any apparently extravascular blood in the brain or within the cranium that was associated with clinical deterioration, as defined by an increase of 4 points or more in the score on the NIHSS, or that led to death and that was identified as the predominant cause of the neurological deterioration.
Hemorrhage in other parts | 36 hours after thrombolysis
  The proportion of patients with other bleeding events was defined by GUSTO bleeding at 90 days
Mortality at 90 days | 90 days after thrombolysis
  Mortality of all-cause

CONTACTS AND LOCATIONS:
Overall Officials: Yunyun Xiong, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Yunyun Xiong, Beijing, China